CLINICAL TRIAL: NCT02246400
Title: CardioMetabolic Program Meets eHealth: Redesign and Evaluation for Optimal Reach and Impact
Acronym: eCMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: # 14-01-290
Record Dates: First submitted 2014-03-18; First posted 2014-09-22 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Obesity; Metabolic Syndrome; Pre-diabetes; Type 2 Diabetes; Cardiovascular Disease
Keywords: eCMP; eHealth; mHealth; Lifestyle intervention; Cardiometabolic risk reduction; PAMF
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Glucose Intolerance; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Intervention (Active Comparator): Usual care for first three months. Initiation of the eCMP after the 3-month time point.
  Interventions: Behavioral: eCMP
- Immediate Intervention (Experimental): Initiation of the eCMP immediately upon completion of baseline data collection and randomization
  Interventions: Behavioral: eCMP

INTERVENTIONS:
Behavioral: eCMP — eCMP is a 6-month lifestyle intervention designed and led by a team of experienced health professionals, including physicians, researchers, dietitians, and registered nurses. The program consists of weekly home and class activities delivered through online or take-home videos, video conferencing, and/or in-person sessions.
  Other Names: Electronically-mediated CardioMetabolic Program (eCMP)

SUMMARY:
The eCMP Pilot aims to study the feasibility and potential effectiveness of an electronically-mediated CardioMetabolic Program (eCMP) for therapeutic lifestyle change among adults with or at high risk for type 2 diabetes, heart disease, and/or stroke.

DETAILED DESCRIPTION:
The eCMP is an evidence-based lifestyle intervention using a holistic, mind-body-spirit-based, and multidisciplinary approach, and it will be delivered using existing web and mobile technologies. In this pragmatic randomized controlled trial, participants will be recruited from primary care patients of an integrated ambulatory care system. They will be randomly assigned to receive the eCMP upon completion of baseline data collection (the Immediate Intervention group) or after 3 months (the Delayed Intervention group). All participants will be assessed at 0, 3 and 6 months. Outcomes include common cardiometabolic risk factors (e.g., weight, blood pressure, and fasting plasma glucose), health behaviors (e.g., dietary intake and physical activity), and indicators of eCMP engagement and adherence (e.g., attendance and self-monitoring).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults aged 18+ years
* High-risk primary prevention: BMI 35+ and prediabetes (including hx of gestational diabetes) and/or metabolic syndrome
* Secondary prevention: BMI 30+ and type 2 diabetes and/or cardiovascular disease
* Able and willing to provide written informed consent

Exclusion Criteria:

* Medical determination that the study is inappropriate or unsafe for the patient
* Type 1 diabetes
* Safety concerns related to significant physical or mental health issues or life expectancy of less than 12 months
* Currently pregnant or lactating
* No regular telephone or broadband Internet access or otherwise unable to participate in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in measure of Health-related quality of life from baseline to 6-months follow up. | 6-months
  SF-8 questionnaire

SECONDARY OUTCOMES:
Change in composite measure of Metabolic Syndrome | 6-months.
  Composite measure of Metabolic Syndrome (criterion factors: waist circumference, blood pressure, fasting plasma glucose, triglycerides, High-density lipoprotein, and body mass index.)
Dietary Intake | Baseline, 3-months, and 6-months.
  Nutrition Data System for Research (NDSR).
Physical Activity | Baseline, 3-months, and 6-months.
  Seven-Day Physical Activity Recall (PAR).
Intervention adherence | 3-months and 6-months.
  Intervention session attendance of virtual classes and in-person physical activity classes.
Body weight | Baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — Palo Alto Medical Foundation; Tak Poon, MD, PharmD, ABIHM, FACC, Principal Investigator — Palo Alto Medical Foundation
Locations (1):
- Palo Alto Medical Foundation, Mills Peninsula Division, Burlingame, California, United States

REFERENCES:
- [Derived] Azar KM, Koliwad S, Poon T, Xiao L, Lv N, Griggs R, Ma J. The Electronic CardioMetabolic Program (eCMP) for Patients With Cardiometabolic Risk: A Randomized Controlled Trial. J Med Internet Res. 2016 May 27;18(5):e134. doi: 10.2196/jmir.5143. PMID 27234480